CLINICAL TRIAL: NCT02440750
Title: Endometrial Preparation Before Operative Hysteroscopy in Premenopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYSTERO
Record Dates: First submitted 2015-03-18; First posted 2015-05-12 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — dienogest; ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dienogest (Experimental): Women selected for operative hysteroscopy that received for 21 days dienogest 2 mg/die
  Interventions: Procedure: operative hysteroscopy; Drug: Dienogest
- Ulipristal acetate (Experimental): Women selected for operative hysteroscopy that received for 21 days ulipristal acetate 5 mg/die
  Interventions: Procedure: operative hysteroscopy; Drug: Ulipristal acetate

INTERVENTIONS:
Procedure: operative hysteroscopy — Performed under general or local anesthesia, antibioprophylaxis may be administered. Cervical dilatation, will be made in order to introduce the hysteroscope. Operative hysteroscope used will include a handle. The distension of the uterine cavity will be performed with physiological saline or glycocoll, depending on the polarity of the high frequency generator necessary for resection system (monopolar or bipolar), with a pressure of maximum irrigation of 110 mm Hg.
Drug: Dienogest — 21 days administration of dienogest 2 mg/die
  Other Names: Visanne
  Arms: Dienogest
Drug: Ulipristal acetate — 21 days administration of ulipristal acetate 5 mg/die
  Other Names: Esmya
  Arms: Ulipristal acetate

SUMMARY:
The presence of a thin endometrium has an important role in allowing the best conditions for hysteroscopic surgery. The aim of this study is to evaluate the efficacy of a 21 day administration of 2 mg of dienogest versus ulipristal acetate 5 mg, in rapid endometrial preparation to operative hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis at office hysteroscopy of symptomatic submucous myomas with intramural development (G1 and G2)

Exclusion Criteria:

* pregnancy
* other hormonal therapy in the previous 8 weeks
* hepatic or renal impairment
* any medical condition that would increase the surgical risk
* refusal or unable to sign written consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | Change in mm from baseline after farmacological therapy
  We perform a transvaginal ultrasound (baseline) and we measure the maximum thickness of endometrial line; at the time of surgery (operative hysteroscopy) we repeat the ultrasound after pharmacological treatment. It will be expressed in mm

SECONDARY OUTCOMES:
Ovarian follicle dimensions | Change in mm from baseline after farmacological therapy
  We perform a transvaginal ultrasound (baseline) and we measure the maximum diameter of follicles; at the time of surgery (operative hysteroscopy) we repeat the ultrasound after pharmacological treatment. It will be expressed in mm
Endometrial appearance | Change from baseline after farmacological therapy
  We perform a diagnostic hysteroscopy (baseline) and we describe the endometrial appearance; at the time of surgery (operative hysteroscopy) we describe the endometrial appearance after pharmacological treatment
Operative time | Within 2 hours after the end of the hysteroscopy
  It will be expressed in minutes